CLINICAL TRIAL: NCT05176184
Title: A Deep Learning Method to Predict Difficult Laryngoscopy Using Cervical Spine X-ray Image: Prospective Validation Study
Brief Title: A Deep Learning Method to Predict Difficult Laryngoscopy Using Cervical Spine X-ray Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2111-111-1272
Record Dates: First submitted 2021-12-12; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Thyroid; Surgery; Intubation; Difficult or Failed
Keywords: deep learning; cervical spine X-ray; difficult laryngoscopy
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: A deep learning model for predicting a difficult laryngoscopy based on a cervical spine lateral X-ray image — The deep learning model uses the input of preprocessed C-spine lateral X-ray images and outputs the level of difficulty of a laryngoscopy. The easy laryngoscopy is defined as a combination of the Cormack-Lehane grades 1-2 and the difficult laryngoscopy is defined as a combination of grades 3-4.
  In addition, before general anesthesia, airway evaluations related to the difficulty of laryngoscopy are performed and the results are compared with the actual level of difficulty.

SUMMARY:
An unanticipated difficult laryngoscopy is associated with serious airway-related complications. The investigators developed a deep learning-based model that predicts a difficult laryngoscopy (Cormack-Lehane grade 3-4) from a cervical spine lateral X-ray using data from 14,135 patients undergoing thyroid surgery. This model showed excellent predictive performance, which was higher than that of other deep learning architectures. In this study, the investigators prospectively validate the model for predicting a difficult laryngoscopy and compare predictive power with clinical airway evaluation.

DETAILED DESCRIPTION:
Predicting a difficulty of a laryngoscopy is important for patient safety, as an unanticipated difficult laryngoscopy is associated with serious airway-related complications, such as brain damage, cardiopulmonary arrest, or death. Although clinical predictors, such as the modified Mallampati classification, thyromental distance, inter-incisor gap, and the upper lip bite test, are used for airway evaluation in clinical practice, these indicators have low sensitivity and large inter-assessor variability and require patient cooperation.

The investigators developed a deep learning-based model that predicts a difficult laryngoscopy from a cervical spine lateral X-ray using data from 14,135 patients undergoing thyroid surgery. And this study is under submission.

This deep learning model showed the highest performance in predicting difficult laryngoscopy compared to other deep learning models (VGG-Net, ResNet, Xception, ResNext, DenseNet, and SENet) with a sensitivity of 95.6%, a specificity of 91.2%, and an area under ROC curve (AUROC) of 0.972.

However, as the model was a retrospective design using existing medical records, the presence or absence of cricoid pressure to obtain the optimal laryngoscopy was not evaluated, and not compared with airway evaluations.

In this study, the investigators prospectively validate the model for predicting a difficult laryngoscopy and compare predictive power with clinical airway evaluation. If this study prospective confirm our results, this approach can be helpful in improving patient safety and preventing airway-related complications through objective and accurate airway evaluation.

ELIGIBILITY:
Inclusion Criteria:

* elective thyroid surgery under general anesthesia

Exclusion Criteria:

* age < 18 years
* no C-spine lateral X-ray image obtained within 3 months before surgery
* Patient who safety is not guaranteed when using a direct laryngoscope. (poor dental condition, risk of neck extension)
* Patients who not cooperate with the physical examination for airway evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergoing thyroid surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 367 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
The area under the receiver operating characteristic curve of deep learning model and airway evaluations for predicting a difficult laryngoscopy. | during induction of anesthesia
  Difficult laryngoscopy definition: Cormack-Lehane grade 3 or 4 . Airway evaluations: Inter-incisor gap (millimeter), thyromental distance (millimeter), thyromental height (millimeter), sternomental distance (millimeter), and modified Mallampati class

SECONDARY OUTCOMES:
The area under the receiver operating characteristic curve of deep learning model and airway evaluations for predicting a difficult intubation. | during induction of anesthesia
  Difficult intubation: Intubation Difficulty Scale (score)
Other Performances for predicting a difficult laryngoscopy of deep learning model. | during induction of anesthesia
  sensitivity (percent), specificity(percent), Positive predictive value(percent), Negative predictive value (percent), F1-score, and balanced accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Chul Lee, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Select A State Or Province, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook TM, MacDougall-Davis SR. Complications and failure of airway management. Br J Anaesth. 2012 Dec;109 Suppl 1:i68-i85. doi: 10.1093/bja/aes393. PMID 23242753
- [Background] Lundstrom LH, Vester-Andersen M, Moller AM, Charuluxananan S, L'hermite J, Wetterslev J; Danish Anaesthesia Database. Poor prognostic value of the modified Mallampati score: a meta-analysis involving 177 088 patients. Br J Anaesth. 2011 Nov;107(5):659-67. doi: 10.1093/bja/aer292. Epub 2011 Sep 26. PMID 21948956
- [Background] De Cassai A, Boscolo A, Rose K, Carron M, Navalesi P. Predictive parameters of difficult intubation in thyroid surgery: a meta-analysis. Minerva Anestesiol. 2020 Mar;86(3):317-326. doi: 10.23736/S0375-9393.19.14127-2. Epub 2020 Jan 8. PMID 31922378
- See also: VGG-Net — https://arxiv.org/abs/1409.1556
- See also: ResNet — https://ieeexplore.ieee.org/document/7780459
- See also: Xception — https://ieeexplore.ieee.org/document/8099678
- See also: ResNext — https://ieeexplore.ieee.org/document/8100117
- See also: DenseNet — https://ieeexplore.ieee.org/document/8099726
- See also: SENet — https://arxiv.org/abs/1709.01507